CLINICAL TRIAL: NCT06014879
Title: Strengths-Based Multi-Level Behavioral Intervention to Promote Resilience and Self-Management in Youth With Type 1 Diabetes
Brief Title: EMPoWER Study - Strengths-based Behavioral Intervention for Youth With Type 1 Diabetes
Acronym: EMPoWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Marisa Hilliard, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-51765
Record Dates: First submitted 2023-08-16; First posted 2023-08-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; youth; adolescent; child; positive psychology; mhealth; ehealth
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: For the first phase of this project, all teen participants (up to 40 total) will create videos about living well with type 1 diabetes. The videos will be used in the upcoming randomized clinical trial of the new intervention.
  For the randomized control trial, a parallel two group design will be used to evaluate the intervention among n=250 parents and youth dyads assigned to the Type 1 Doing Well intervention condition or the enhanced usual care condition (1:1). All parent and youth dyads are randomized to either the Type 1 Doing Well intervention condition or the enhanced usual care condition. Parents and youth dyads will be in the the study for approximately 12 months.
  Providers (up to 20 per site, 40 total) will also be enrolled as participants to deliver the provider conversation intervention to parent and youth dyads randomized to the intervention condition, and to provide data about their experiences.
Masking Description: For the randomized control trial, because of the nature of the behavioral intervention, participants and investigators will be aware of their assignment to the intervention condition or the enhanced usual care condition.
  For the teen videos, all video participants will be in a single group, so there will be no masking. For diabetes care professionals, all participants will be in a single group, so there will be no masking. Teen video participants and diabetes care professional participants will not receive interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Type 1 Doing Well (T1DW) Program (Experimental): Youth with type 1 diabetes (ages 10-13) and their parents or legal guardians who are receiving care from enrolled diabetes care providers will be randomized to either the T1DW Program or the EUC Program. After being randomized to the T1DW Program at the orientation session, parents and youth will receive an overview of the web-based mobile application and intervention activities that they will engage with for 6 months. The app-based intervention activities include brief daily use of the app for parents to recognize and reinforce their child's positive diabetes-related behaviors, brief weekly activities for parents and youth to reflect on and discuss what the child has done well for diabetes, family diabetes goal-setting, and videos for parents and youth about living well with T1D. Parents and youth will also engage in a brief strengths-based conversation with their diabetes care provider at one medical appointment during the study period.
  Interventions: Behavioral: Type 1 Doing Well (T1DW) Program
- Diabetes-Related Information and Resources Program (Enhanced Usual Care; EUC) (Active Comparator): Youth with type 1 diabetes (ages 10-13) and their parents or legal guardians who are receiving care from enrolled diabetes care providers will be randomized to either the T1DW Program or the EUC Program. After being randomized to the EUC Program at the orientation session, parents and youth will receive monthly email handouts with diabetes-related information and resources for 6 months.
  Interventions: Other: Diabetes-Related Information and Resources Program

INTERVENTIONS:
Behavioral: Type 1 Doing Well (T1DW) Program — Parent and youth will each have access to a version of the app. The study app activities include parents and youth:
  * noticing what the youth does well for diabetes;
  * setting and tracking a family diabetes goal in the app; and
  * having a weekly meeting to review what the youth is doing well with diabetes and progress on the family diabetes goal.
  Parents and youth will also have access to age-appropriate libraries of videos with diabetes-specific content.
  Parents and youth will also have a conversation with the youth's diabetes care provider at a regularly scheduled diabetes appointment at participating hospital sites.
  Arms: Type 1 Doing Well (T1DW) Program
Other: Diabetes-Related Information and Resources Program — Parent and youth will receive diabetes-related information and resources in the form of electronic handouts. They will receive one handout per month by email during the 6-month intervention period. These handouts include a variety of diabetes-related topics curated by the study team. Handouts will not include any specific information about the youth's health.
  Other Names: Enhanced Usual Care (EUC) Program
  Arms: Diabetes-Related Information and Resources Program (Enhanced Usual Care; EUC)

SUMMARY:
The EMPoWER Study randomized clinical trial is a strengths-based behavioral intervention delivered to youth with type 1 diabetes (age 10 to 13) and their parents. The purpose of the intervention is to improve glycemic, behavioral, and psychosocial outcomes in youth with diabetes using a multiple systems approach that engages youth, their parents, and diabetes care providers to identify and build youths' diabetes strengths. The primary aim of this study is to assess the intervention impact on glycemic control, adherence, and health-related quality of life (HRQOL). Secondary aims are to evaluate behavioral mediators of intervention impact and to examine intervention dose as a mediator of intervention impact.

DETAILED DESCRIPTION:
The goal of the randomized clinical trial (RCT) is to learn if a brief behavioral intervention targeting multiple systems ("Type 1 Doing Well" Program) can improve glycemic, behavioral, and psychosocial outcomes in youth with type 1 diabetes. Youth, age 10 to 13, will enroll with one parent or legal guardian to participate in the study with them. Researchers will compare the Type 1 Doing Well (T1DW) Program arm to the Enhanced Usual Care (EUC; "Diabetes-Related Information and Resources" Program) arm.

Parent-youth dyads in both study arms will provide data (e.g. questionnaires, A1c, medical chart and diabetes device data) at four timepoints throughout the duration of the study. Following baseline data collection, parent-youth dyads will complete an orientation session with study team members to be randomized to their study arm and review study activities. Parent and youth will also be invited to complete a feedback interview on their experience with the program they received.

The intervention will take place during the 6-month intervention period, and participants will be randomly allocated to 1 of two intervention conditions:

1. Parents and youth in the T1DW Program condition (intervention) will use a web-based mobile application to do daily and weekly activities focused on recognizing and reinforcing youths' diabetes strengths. They will also have a conversation with the youth's diabetes provider about what is going well in diabetes care at a routine diabetes appointment.
2. Parents and youth in the EUC Program condition will receive and review 6 monthly diabetes-related information and resources in the form of electronic handouts.

In preparation for the randomized clinical trial of a new behavioral intervention for preteens with type 1 diabetes and their parents, the study is also enrolling adolescents with type 1 diabetes to create videos about living well with type 1 diabetes. The videos will be used in the intervention materials for the randomized clinical trial.

Diabetes care providers at each of the sites will also be enrolled in the study. Provider participants will receive a brief training to deliver the strength-based conversation with parent-youth dyads in the T1DW Program arm, and they will complete study-related questionnaires about their experiences delivering the strengths-based conversation component of the intervention.

ELIGIBILITY:
For Trial Participants -

Inclusion Criteria:

Youth

* type 1 diabetes diagnosis per ADA criteria for at least 6 months,
* age 10 to 13 years at consent,
* English or Spanish fluency,
* At least one hemoglobin A1c value ≥ 8 % (percent) within the past 12 months
* Patient at one of the participating study sites

Parent/legal guardian of youth

* Age at least 18 years old at time of consent,
* English or Spanish fluency,
* Consistent access to a mobile phone that has texting capabilities and a device with internet access

Exclusion Criteria:

Youth

Being treated for:

* a major serious or acute medical condition or comorbidity (e.g. cancer, cystic fibrosis),
* a major serious psychological or psychiatric condition,
* a major serious developmental condition that would interfere with capacity for informed assent or participation or that would confound outcomes

Parents/legal guardian of youth participant

Being treated for:

* a major serious or acute medical condition or comorbidity (e.g. cancer, cystic fibrosis),
* a major serious psychological or psychiatric condition,
* a major serious developmental condition that would interfere with capacity for informed consent or participation or that would confound outcomes

Other Exclusion Criteria

* Plans to move diabetes care out of participating hospital site within next 6 months,
* Legal guardianship of the youth with diabetes being unclear at the time of screening or recruitment,
* Study team learning of other involvement with the legal system during screening or recruitment

For the Teen Videos:

Inclusion Criteria:

* self-reported type 1 diabetes diagnosis for ≥ 1 year,
* age 14-17 at consent,
* English fluency,
* living in the United States

Exclusion Criteria:

* major psychiatric or developmental disorders in youth or parents that would interfere with capacity for informed consent or participation,
* major medical comorbidities that would confound outcomes (e.g., cancer, cystic fibrosis).

Diabetes Care Provider Participants

Inclusion Criteria:

- Provider at one of the sites' diabetes care centers

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic and Medical Information Questionnaire | Baseline
  Only demographic information and limited diabetes treatment information will be collected about participants in the teen videos portion of this study. Participants will complete a brief questionnaire developed by the study team, which will request self-reported information about participant demographics (e.g., race, ethnicity, gender) and medical information (e.g., time since diabetes diagnosis, current treatments).
Glycemic Control - HbA1c | Baseline, 6 months, 12 months
  Point of care HbA1c values documented by the medical team at each clinic visit will be collected from the electronic health record, to assess change in glycemic outcomes. Youth will be asked to complete a home dry blood spot A1c kit at three study timepoints unless an A1c value is documented in the electronic health record within the required timeframe. The study team will mail youth a home kit with instructions, all necessary materials to collect the sample, and a pre-paid mailer to ship it back. Higher HbA1c indicates higher average blood glucose values over the previous 2-3 months, which represents poorer glycemic control.
Glycemic Control - time-in-range | Baseline, 3 months, 6 months, and 12 months
  When available for youth who use a continuous glucose monitor (CGM), 14 days' of CGM data will be downloaded at each time point by the study teams to calculate glucose time-in-range as an additional index of glycemic control. Higher time-in-range is an indicator of better glycemic control.
Adherence - Self-Care Inventory 2 (SCI-2) | Baseline, 3 months, 6 months, and 12 months
  Parents and youth will complete the Self-Care Inventory 2 (SCI-2) Short Form. The form was adapted/shortened by the study team with permission from the original author, with validation paper forthcoming. Higher scores indicate higher adherence/more engagement in diabetes self-management behaviors.
Health-Related Quality of Life (HRQOL) | Baseline, 3 months, 6 months, and 12 months
  Parents and youth willcomplete the age- and respondent-appropriate version of the Type 1 Diabetes and Life (T1DAL) measure. Psychometric data regarding the validity and reliability of the pediatric, adult, and parent/partner versions of the T1DAL are published. Total scores are on a 100-point scale, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Diabetes Distress | Baseline, 3 months, 6 months, and 12 months
  Parents and youth will complete the age- and respondent-appropriate version of the Problem Areas in Diabetes (PAID) scale (children, adolescents, and parents). Higher scores on the measure indicate more distress.
Diabetes Strength | Baseline, 3 months, 6 months, and 12 months
  The Diabetes Strengths and Resilience (DSTAR) measure assesses youths' self-perceptions about what they do well with diabetes (known as diabetes strengths). Youth will rate how often the items represent their experiences/perspectives about their diabetes strengths. Items responses range from 0 (never) to 4 (almost always) and are calculated for total and subscale scores (higher = more strengths).
Positivity Scale | Baseline, 3 months, 6 months, and 12 months
  The Positivity Scale assesses the tendency to view life and experiences with a positive outlook. Parents respond to an 8-item measure on a scale from 1 (Strongly Disagree) to 5 (Strongly Agree) and are calculated for total scores (higher = more positivity).
Role Overload | Baseline, 3 months, 6 months, and 12 months
  The Role Overload questionnaire is a 6-item scale that assess parents' self-perceptions about role overload they are experiencing. Parents indicate how often they feel role overload on a scale from 1 (Never) to 7 (Always) and are calculated for total scores (higher = more role overload).
Family Conflict - Diabetes Family Conflict Scale - Revised (DFCS) | Baseline, 3 months, 6 months, and 12 months
  The Diabetes Family Conflict Scale-Revised (DFCS) is a 19-item scale assessing parent and youth perceptions of disagreements related to diabetes care. This measure has been used extensively with youth with diabetes and parents of youth with diabetes and is valid and reliable.
Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Positive Affect 15a Items | Baseline, 3 months, 6 months, and 12 months
  The PROMIS Short Form Positive Affect 15a assesses momentary positive or rewarding affective experiences. Youth respond to 3 items on a scale from 1 (Never) to 5 (Always) and are calculated into a total score (higher = more positive affect).
PROMIS Short Form Family Relationships 4a Items | Baseline, 3 months, 6 months, and 12 months
  The PROMIS Short Form Family Relationships 4a assesses the subjective (affective, emotional, cognitive) experience of being involved with one's family. Youth respond to 6 items on a scale from 1 (Never) to 5 (Always) and are calculated into a total score (higher = more family support).
Satisfaction Questionnaire | 3 months, 6 months, and 12 months
  Parents and youth will complete a satisfaction survey both post-intervention and at 12-month follow-up to rate their experiences in the study while the intervention group will also rate the usefulness of and their satisfaction with the intervention components mid-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Hilliard, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be available within study team. Participants in the teen videos may be identified by showing face within videos, and participants sign consent form and institutional media release forms.